CLINICAL TRIAL: NCT01721863
Title: Effects of Exercise Training on Endothelial Function, Heart Rate Variability, Exercise Capacity, and Quality of Life in Patients With Permanent Atrial Fibrillation
Brief Title: Effects of Exercise Training in Patients With Permanent Atrial Fibrillation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201010032R
Record Dates: First submitted 2010-11-22; First posted 2012-11-06 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Exercise Training; Endothelial Function; Autonomic Nerve Modulation; Exercise Capacity; Quality of Life
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Exercise group will undergo progressively aerobic exercise training with 40-85% maximal oxygen consumption for 40 minutes, 3 sessions per week for 12 weeks.
  Interventions: Other: Exercise training
- control group (No Intervention): Control group conducted the usual care

INTERVENTIONS:
Other: Exercise training — Exercise group will undergo progressively aerobic exercise training with 40-85% maximal oxygen consumption for 40 minutes, 3 sessions per week for 12 weeks.
  Other Names: Aerobic exercise Training
  Arms: Exercise training

SUMMARY:
Atrial fibrillation (AF) is a common arrhythmia. The proposed patholophysiological mechanisms of AF include abnormal electrical conduction in atrium and sympathovagal imbalance with increased vagal tone. Patients with AF have poor exercise capacity that may contribute to decreased atrial effective refractory period, and decreased cardiac output and heart rate reserve, and may result in poor quality of life. Poor endothelial function had been noted in patients with AF, associated with increased risks of cerebrovascular and cardiovascular disease. Exercise training has been noted to improve exercise capacity and quality of life in patients with AF only in some studies. Endothelial function can be improved by exercise training in patients with cardiovascular disease, but no report in patients with AF. Evidence of exercise training is still needed in patients with AF. The purpose of this study is to investigate the effect of exercise training on

1. endothelial function
2. heart rate variability
3. exercise capacity
4. quality of life.

DETAILED DESCRIPTION:
A randomized controlled study was implemented to examine :(1) the effect of interval aerobic exercise training combined with resistance training on endothelial function, heart rate variability (HRV), exercise capacity, and quality of life (QoL); (2) the influential factors related to exercise capacity, and the relationship between exercise capacity and quality of life in patients with permanent atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial fibrillation≥ 1 year aged 40-76 years
* Recurrence AF after ablation
* Under antiarrhythmia medication control

Exclusion Criteria:

* CAD or myocardial infrarction history
* NYHA≥ III-IV, or LVEF≤45%
* Mitral or aortic valve regurgitation ≥ Gr. II
* Mitral valve or aortic valve stenosis
* Pacemaker
* Cardioversion by ablation
* Pulmonary artery hypertension
* Any surgery in previous 3 months
* Any neurological disorders
* Cancer
* Severe musculoskeletal disorder
* Hyperthyroidism
* Premenopausal women

Ages: 40 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change of exercise capacity (after intervention) | At baseline and 12 weeks after intervention
  To measure maximal oxygen consumption, maximal oxygen pulse, maximal heart rate and blood pressure, cumulated and peak workload by cycle ergometer with Vmax 229 system

SECONDARY OUTCOMES:
Change of heart rate variability (after intervention) | At baseline and 12 weeks after intervention
  To record ECG by lead V1 with KENZ 170 on supine position for 1 hour
Change values of head up tilt test (after intervention) | At baseline and 12 weeks after intervention
  Subjects were tilted up 60 degree on tilting table for 15 minutes to record the change of blood pressure and heart rate, and heart rate variability.
Change of endothelial function (after intervention) | At baseline and 12 weeks after intervention
  To measure dependent-endothelial moulation by flow-mediated dilatation with Sonosite 180 portable ultrasound.
Change of quality of life (after intervention) | At baseline and 12 weeks after intervention
  To measure quality of life by Short-form 36 and symptom checklist

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan